CLINICAL TRIAL: NCT03915470
Title: A Phase 2 Study to Assess the Effect of a Repeated Dose of XF-73 Nasal Gel on the Microbiological Burden of Commensal Staphylococcus Aureus Nasal Carriage in Surgical Patients at Risk of Post-operative Staphylococcal Infections
Brief Title: Effect of Exeporfinium Chloride (XF-73) Gel on Nasal S.Aureus in Patients at Risk of Post-op Staphylococcal Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Destiny Pharma Plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: XF-73B07
Record Dates: First submitted 2019-04-01; First posted 2019-04-16 (Actual); Results first posted 2022-06-01 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2022-05

CONDITIONS: Staphylococcal Infections; Surgical Site Infection
Keywords: Post-operative; Post-surgical; Infection prevention; Staphylococcus aureus; MSSA; MRSA
MeSH Terms: conditions — Staphylococcal Infections; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XF-73 (Experimental): 0.3 mL applications in each naris of 0.2% w/w XF-73 nasal gel for a cumulative dose of 6.0 mg of XF-73.
  Interventions: Drug: XF-73
- Placebo (Placebo Comparator): 0.3 mL applications in each naris of placebo to match XF-73 nasal gel.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XF-73 — XF-73 is a dicationic porphyrin derivative having potent bactericidal properties with a novel mode of action.
  Other Names: Exeporfinium chloride
  Arms: XF-73
Drug: Placebo — Placebo to match XF-73 nasal gel for colour and viscosity.
  Other Names: Matched Placebo
  Arms: Placebo

SUMMARY:
This study looks at the difference between XF-73 and placebo in reducing the carriage of a bacteria S. aureus in the nose before, during and after heart surgery. Only people who normally have S.aureus in their nose will be enrolled onto the study. This will be confirmed by analysis of a nasal swab (a cotton bud placed in the nose) before entering the study. It is expected 125 people will participate in this study. Participation will be confirmed by analysis of a nasal swab (a cotton bud placed in the nose) before entering the study. XF-73 or placebo will be given 5 times, with an equal chance of participants receiving either XF-73 or placebo. During the hospital stay more nasal swabs will be taken to determine the amount of S.aureus present in the participant's nose. Other tests such as blood samples, blood pressure and an examination of the nose and sense of smell will be performed as part of the safety assessment. After the hospital stay participants will be followed up for 30 days or if a device has been inserted into the body as part of the surgery for 90 days to look at the rates of post-operative infection between the placebo and XF-73 groups. The study will run for about 18 months. During this period, an independent data monitoring committee will review the study to make sure that the balance of benefits and risks of participating in the study does not change.

DETAILED DESCRIPTION:
This is a multi-centre, double blind, randomized, placebo-controlled study of multiple applications of a single concentration of XF-73 nasal gel to assess the microbiological effect of XF-73 on commensal S. aureus nasal carriage in patients scheduled for surgical procedures deemed to be at high risk of post-operative S. aureus infection. The study is divided in 4 periods: screening (days -14 to -1) randomization (days -10 to -1), treatment (days -1 and 0) and follow-up (post-last study dose to day 30 or day 90 if an implant is inserted during surgery). Day 0 is the calendar day in which surgery takes place. Only patients who test positive to S. aureus by a centrally-performed rapid diagnostic test will be enrolled in the study. Approximately 125 patients will be randomly allocated in a 1:1 ratio to 0.2% w/w XF-73 nasal gel treatment OR placebo to match XF-73 nasal gel.

The study drug, 0.2% w/w XF-73, or matched placebo will be administered 4 times into each nostril over 24 hours prior to surgery and then a single application immediately upon closure of surgical wound. Additionally, patients may undergo chlorhexidine skin decolonisation ahead of surgery and receive perioperative prophylactic systemic antibiotics in accordance with local practice.

Efficacy will be assessed by S. aureus colonisation from screening to 7 days after surgery as well as by incidence of post-operative staphylococcal infections and use of anti-staphylococcal antibiotics post-surgery. Safety will be assessed by reported adverse events (AEs) from screening up to Day 7 as well as vital signs, physical examination (ENT), clinical laboratory assessments (haematology, clinical chemistry, and urinalysis) and Smell Identification Tests at different time points throughout the study.

The maximum study duration will be 45 or 105 days for each individual (from screening to post-study follow-up visit) depending on whether a foreign implant was inserted during surgery.

An independent data monitoring committee (IDMC) will be set up which will review the safety information from the study, the incidence of post-operative staphylococcal infections and to ensure that the balance of benefits and risks of participating in the study does not change.

ELIGIBILITY:
Individuals who meet all of the following criteria are eligible to participate in the study.

1. Male or female patients between 18 and 75 years of age.
2. Patients who are confirmed nasal S. aureus carriers by polymerase chain reaction (PCR) screen assay, and due to undergo surgical procedure.
3. Patients who are willing to provide written informed consent.
4. Patients who are willing and able (as per Investigator judgment) to complete all protocol specified visits and assessments.
5. Woman of childbearing potential* with a negative urine pregnancy test (sensitive to 25 IU human chorionic gonadotropin (hCG)).

   * Women of childbearing potential are defined as those women between menarche and menopause who have not undergone permanent sterilisation. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy, and bilateral oophorectomy.

Individuals who meet any of the following criteria are not eligible to participate in the study.

1. Pregnancy (current) or currently lactating.
2. Uncontrolled acute or chronic illness (as determined by the investigator) in addition to those requiring the planned surgical intervention.
3. History of atopy, allergic reactions or hypersensitivity to the study medication or its components.
4. Current upper respiratory tract infection, cold or influenza with significant nasal symptoms that might impact on the patient's ability to comply with the gel application procedure.
5. History of photosensitivity.
6. Family history of porphyria.
7. Use of intra-nasal topical or systemic antibiotics or anti-infectives within the last 4 weeks before screening. (Patients who screen positive for nasal carriage of S. aureus and receive topical or systemic antibiotics or anti-infectives which are not part of their prophylactic peri-operative SOC between screening and first dose of investigational medicinal product (IMP) will be excluded from the study.) The use of intra-nasal antibiotics or anti-infectives other than the study medication prior to surgery is not allowed.
8. Use of other prescribed or over the counter nasal medication in the last 14 days, or oral decongestants in the last 7 days before first administration of study drug.
9. Participation in a clinical trial within the last 12 weeks before first administration of study drug.
10. Contemporaneous clinically significant abnormalities in vital signs or laboratory analyses reported within 14 days prior to randomization which in the opinion of the Investigator would preclude from the safety assessment of the medication under study.
11. Nasal polyps or significant anatomical or other nasal abnormality that would prevent from appropriate administration of the study treatment or represent an excessive risk for the patient's participation.
12. History of nasal surgery including cauterization.
13. A recent history of frequent epistaxis and/or an episode of epistaxis within 3 months of the planned surgery.
14. Use of in situ nasal jewellery or existence of open nasal piercings.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2019-08-29 (Actual); Primary Completion 2021-01-04 (Actual); Study Completion 2021-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jesus M Gonzalez Moreno, MD, Study Chair — Destiny Pharma Plc; Jim P Lees, BSc, Study Director — Destiny Pharma Plc
Locations (21):
- United States (7):
  - University of Florida, Gainesville, Florida
  - Snake River Research, PLLC, Pocatello, Idaho
  - MercyOne Iowa Heart Center, Des Moines, Iowa
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - University of Missouri Health Care, Columbia, Missouri
  - Memorial Hermann - Memorial City Medical Center, Houston, Texas
  - CHI Franciscan Research Center, Tacoma, Washington
- Georgia (10):
  - Ltd Clinic LJ, Kutaisi
  - Ltd Israel-Georgia Medical Research Clinic Helsicore, Tbilisi
  - Ltd "Open Heart", Tbilisi
  - Ltd Cardiology Clinic Guli, Tbilisi
  - Ltd Acad. G.Chapidze Emergency Cardiology Center, Tbilisi
  - Ltd Bokhua Memorial Cardiovascular Center, Tbilisi
  - Ltd Tbilisi Heart and Vascular Clinic, Tbilisi
  - Ltd Clinic Jerarsi, Tbilisi
  - Ltd Tbilisi Heart Center, Tbilisi
  - JSC Evex Hospitals, Tbilisi
- Serbia (4):
  - Clinical Center of Serbia, Belgrade
  - Clinic for Cardiac Surgery, Institute for Cardiovascular Disease-Deinje, Belgrade
  - Institute for Cardiovascular Disease of Vojvodina, Kamenitz
  - Clinical Center Nis, Niš

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Mangino JE, Firstenberg MS, Milewski RKC, Rhys-Williams W, Lees JP, Dane A, Love WG, Gonzalez Moreno J. Exeporfinium chloride (XF-73) nasal gel dosed over 24 hours prior to surgery significantly reduced Staphylococcus aureus nasal carriage in cardiac surgery patients: Safety and efficacy results from a randomized placebo-controlled phase 2 study. Infect Control Hosp Epidemiol. 2023 Jul;44(7):1171-1173. doi: 10.1017/ice.2023.17. Epub 2023 Mar 23. PMID 36951472

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants at risk of post surgery staphylococcal infections were recruited based on physician assessment across 20 sites (14 enrolling) between June 2019 and March 2021. The first participant was enrolled on 29 August 2019 and the last participant was enrolled on 29 December 2020.
Pre-assignment Details: 124 enrolled participants
Groups:
- XF-73: Participants received 0.3 mL applications in each naris of 0.2% w/w XF-73 nasal gel 4 times in one day prior to surgery and once more after surgery, for a cumulative dose of 6.0 mg of XF-73.
- Placebo: Participants received 0.3 mL applications in each naris of placebo to match XF-73 nasal gel, 4 times in one day prior to surgery and once more after surgery.
  Note: Placebo to match XF-73 nasal gel for colour and viscosity.
Period: Overall Study
Arm/Group | XF-73 | Placebo
Started | 63 | 61
Completed | 57 (63 - 6 (discontinued intervention)) | 59 (61-2 (discontinued intervention))
Not Completed | 6 | 2
Not completed — Death | 3 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — XF-73: Failure to meet RND criteria, Placebo: Surgery was cancelled | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all patients who received at least 1 dose of study drug
Groups:
- Total: Total of all reporting groups
Arm/Group | XF-73 | Placebo | Total
Number analyzed (Participants) | 63 | 61 | 124
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.5 (9.93) | 61.2 (8.79) | 60.9 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 30
  Male | 46 | 48 | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 3 | 4
  Not Hispanic or Latino | 59 | 56 | 115
  Unknown or Not Reported | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 63 | 61 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 2 | 6
  Georgia | 55 | 56 | 111
  Serbia | 4 | 3 | 7
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — units: kg/m2 Mean (Standard Deviation) Population: Intent-To-Treat Population Set
  kg/m^2
    number analyzed (Participants) | 62 | 59 | 121
    (all) | 30.410 (4.4140) | 30.055 (4.7368) | 30.237 (4.5586)

OUTCOME MEASURES:

1. Primary Outcome: Change in S. Aureus Log CFU/mL From Baseline to Pre-surgery
Description: To demonstrate the efficacy of a 0.2% XF-73 nasal gel in reducing the microbiological burden of nasal S. aureus measured as change in colony forming units (CFU) per millilitre (mL) from baseline to immediately prior to surgery in a patient population at risk of post-operative staphylococcal infection
Time Frame: Baseline (Day-10 to Day-1) to immediately prior to surgery (Day 0)
Population: microbiological Intent-To-Treat (micro ITT) set: all patients who were randomized, received at least 1 dose of study drug, have at least 1 post-baseline assessment of S. aureus log10 CFU/mL and who have a log10 CFU/mL result at baseline greater than 0, i.e. all patients in the mITT set with a quantifiable baseline microbiological result.
Measure: Mean (Standard Deviation); unit: log10 (CFU/mL)
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 43 | 40
log10 (CFU/mL) | -2.842 (1.8552) | -0.469 (1.3697)

2. Secondary Outcome: Change in S. Aureus Log CFU/mL From Baseline to Immediately Post-surgery
Description: To determine the effect of a 0.2% XF-73 nasal gel on S. aureus nasal burden measured as CFUs/mL in follow-up after last administration.
Time Frame: From baseline (day -10 to Day -1) to immediately post surgery (Day 0)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 (CFU/mL)
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 43 | 40
log10 (CFU/mL) | -2.773 (1.8531) | -0.314 (1.7674)

3. Secondary Outcome: Change in S. Aureus Log CFU/mL From Baseline to 48 Hours After Surgery
Description: To determine the effect of a 0.2% XF-73 nasal gel on S. aureus nasal burden measured as CFUs/mL in follow-up 48 hours after last administration.
Time Frame: From baseline to follow-up at 48 hours after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 (CFU/mL)
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 43 | 40
log10 (CFU/mL) | -2.700 (1.7362) | -1.477 (1.6222)

4. Secondary Outcome: Change in S. Aureus Log CFU/mL From Baseline to Immediately After Surgery to 6 Days (± 24hours) After Surgery
Description: To determine the effect of a 0.2% XF-73 nasal gel on S. aureus nasal burden measured as CFUs/mL in follow-up 7 days after last administration.
Time Frame: From baseline to follow-up Day 6 ± 24hours after surgery
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: log10 (CFU/mL)
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 43 | 40
log10 (CFU/mL) | -3.106 (1.7995) | -2.399 (1.6933)

5. Secondary Outcome: Number of Participants With Staphylococcal Post-operative Infections During the 30-day Period After Surgery (90 Days in the Case of Foreign Implant)
Description: To assess the effect of XF-73 on S. aureus nasal carriage in the prevention of post-operative staphylococcal infections (surgical site infection, blood stream infections, and others) during the 30 days post-surgery (90 days in the case of a foreign implant).
Time Frame: From immediately post-surgery to 30 days post surgery (90 days in the case of foreign implant)
Population: Number of microITT patients with post-operative S.aureus infections
  microbiological Intent-To-Treat (micro ITT) set: all patients who were randomized, received at least 1 dose of study drug, have at least 1 post-baseline assessment of S. aureus log10 CFU/mL and who have a log10 CFU/mL result at baseline greater than 0, i.e. all patients in the mITT set with a quantifiable baseline microbiological result.
Measure: Number; unit: participants
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 43 | 40
participants | 0 | 0

6. Secondary Outcome: Incidence of Treatment-emergent Adverse Events From the First Dose of Study Medication to 6 Days (± 24hours) After Last Dose of Study Medication.
Description: To describe the safety and tolerability of multiple administrations of a 0.2% XF-73 nasal gel in a population of surgical patients at risk of post-operative staphylococcal infections.
Time Frame: Immediately prior to surgery until Day 6 ± 24hours.
Population: Total number of TEAEs in the safety set
  Safety set: all patients who received at least 1 dose of study treatment
Measure: Number; unit: events
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 63 | 61
events | 67 | 68

7. Secondary Outcome: Changes in Nasal Examination.
Description: To describe the safety and tolerability of multiple administrations of a 0.2% XF-73 nasal gel in a population of surgical patients at risk of post-operative staphylococcal infections by comparison of changes in ENT specialist nasal examination findings from randomisation to 48hours ± 24hours post surgery.
Time Frame: From Randomisation (Day -10 to Day -1) until 48hours ± 24hours post surgery.
Population: Number of patients in the safety set with clinically significant changes in nasal examination at 48h ± 24h
  Safety set: all patients who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 63 | 61
Participants | 0 | 0

8. Secondary Outcome: Changes in Brief Smell Identification Test (B-SIT).
Description: To describe the safety and tolerability of multiple administrations of a 0.2% XF-73 nasal gel in a population of surgical patients at risk of post-operative staphylococcal infections by comparison of Brief Smell Identification Test (B-SIT) score, assessment and percentile ranking changes from prior to first dose until Day 6 ±24h post surgery.
  Patients are asked to identify 12 unique smells; the more smells they identify correctly the higher the score (0-12). Comparison of the individual patient score is then made against their expected percentile ranking dependent on age and sex of the general population to determine if their percentile ranking is normal, abnormal relative to age or deficit relative to younger persons.
Time Frame: From Randomisation (Day -10 to Day -1) until Day 6 ± 24hours post surgery
Population: Safety set: all patients who received at least 1 dose of study drug
Measure: Count of Participants; unit: Participants
Arm/Group | XF-73 | Placebo
Number analyzed (Participants) | 63 | 61
Participants
  Assessed as 'Normal' at Day 6 ±24h post surgery | 52 | 50
  Assessed as 'Deficit relative to younger persons' at Day 6 ±24h post surgery | 4 | 5
  Assessed as 'Abnormal relative to age' at Day 6 ±24h post surgery | 2 | 1
  Assessed as 'Below percentile rank' at Day 6 ±24h post surgery | 0 | 0
  Assessed as 'Not Done' at Day 6 ±24h post surgery | 0 | 3
  Participants did not complete | 5 | 2

ADVERSE EVENTS:
Time Frame: From screening until 7 days after a subject received first dose
Description: Non-treatment emergent AEs: recorded from the time when the patient is enrolled into the study until first administration of study drug, TEAEs: First Administration of Study Drug to Patient's Day 6 visit,
  Only AEs that meet SAE criteria and are considered related with the study medication by the investigator will be recorded after Day 6 through the final follow up visit
Arm/Group | XF-73 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/63 | 1/61
Serious Adverse Events (participants affected / at risk) | 4/63 | 5/61
Other Adverse Events (participants affected / at risk) | 31/63 | 15/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XF-73 (N=63) | Placebo (N=61)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 1 (1) | 1 (1)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Asymptomatic COVID-19 (Infections and infestations) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | XF-73 (N=63) | Placebo (N=61)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 14 (14)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Pericardial effusion (Cardiac disorders) | 5 (5) | 5 (5)
Atrial Fibrillation (Cardiac disorders) | 5 (5) | 4 (6)

LIMITATIONS AND CAVEATS:
Study recruitment was affected by the impact of the COVID-19 pandemic as hospitals and staff were reassigned to provide care needed to treat patients with COVID-19.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Protocol limits Investigators to not publish any data (poster, abstract, paper, etc.) without having consulted with the Sponsor in advance.

DOCUMENTS (2):
  • Study Protocol (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/70/NCT03915470/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-02): https://cdn.clinicaltrials.gov/large-docs/70/NCT03915470/SAP_001.pdf